CLINICAL TRIAL: NCT03512340
Title: A Phase 1 Study of SRF231 in Patients With Advanced Solid and Hematologic Cancers
Brief Title: Study of SRF231 in Patients With Advanced Solid and Hematologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Surface Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRF231-101
Record Dates: First submitted 2018-03-13; First posted 2018-04-30 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Advanced Solid Cancers; Hematologic Cancers
Keywords: CD47; SiRP α; tumor microenvironment; macrophage; solid tumor; Phase 1; safety; efficacy; hematologic malignancies; SRF231
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: This Phase 1/1b, open-label, first-in-human, monotherapy study will be conducted in 2 parts. Part A will consist of the SRF231 monotherapy dose-escalation portion of the study, and will enroll up to 48 patients with advanced solid tumors and lymphoma/CLL.
  Part B will include 5 monotherapy expansion cohorts: in advance solid and hematologic cancers (100 patients total).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of SRF231 as a monotherapy in patients with advanced solid tumors and lymphoma/Chronic lymphocytic leukemia.
  Interventions: Drug: SRF231
- Part B Cohort 1 (Experimental): Depending upon the results from Part A of the study and the decision from the Safety Review Committee, 1 or 2 doses or dosing frequencies of SRF231 in select advanced solid and hematologic malignancies.
  Interventions: Drug: SRF231

INTERVENTIONS:
Drug: SRF231 — SRF231 specifically blocks the interaction between CD47 and signal regulatory protein alpha and acts as a potent enhancer of human tumor cell phagocytosis.

SUMMARY:
This Phase 1/1b, open-label, first-in-human, monotherapy study will be conducted in 2 parts. Part A will consist of the SRF231 monotherapy dose-escalation portion of the study, and will enroll up to 48 patients with advanced solid tumors and hematological cancers. Part B will include monotherapy expansion cohorts in advanced solid and hematologic cancers to further examine SRF231 as monotherapy (100 patients total).

DETAILED DESCRIPTION:
This first-in-human study is designed to evaluate the safety and tolerability of SRF231 as a monotherapy via dose escalation (Part A), and to determine the dose(s) of SRF231 to be further examined in expansion cohorts as monotherapy. The preliminary clinical activity of SRF231 administered as monotherapy will be characterized, along with pharmacokinetics (PK) and pharmacodynamics. In Part B, the safety and tolerability of SRF231 as monotherapy will be evaluated in select patient cohorts of advanced cancers and evaluate clinical activity. The study also is designed to examine the effect of SRF231 monotherapy on peripheral blood immune cell subsets, peripheral blood gene expression, and serum biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Failure to respond to standard therapy, and for whom no appropriate therapies are available (based on the judgment of the Investigator).
3. Histological or cytological evidence of advanced, relapsed, or refractory, solid and hematologic cancers that are not a candidate for curative therapy.
4. Part B only: Patient must have demonstrated progressive disease (PD) after the most recent treatment regimen (or within 3 months prior to enrollment in the case of treatment-naïve patients).
5. Washout period from the last dose of previous anticancer therapy (chemotherapy, biologic, or other investigational agent) to the initiation of study drug must be > 5 times the half-life of the agent or > 21 days (whichever is shorter).

   Note: the washout period for palliative radiotherapy is 7 days.
6. Resolution of adverse events (AEs) related to prior anticancer therapy (including immune-related AEs but excluding alopecia) to ≤ Grade 1 per NCI-CTCAE v. 4.03 or higher.
7. Measurable disease per applicable disease-specific criteria for Part B only.
8. Serum creatinine clearance ≥ 60 mL/min per Cockcroft-Gault formula or serum creatinine ≤ 2.0 x the upper limit of normal (ULN).
9. Total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN if elevated due to Gilbert's syndrome).
10. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 2.5 x ULN ( < 5 x ULN if liver metastasis).
11. Adequate hematologic function, defined as absolute neutrophil count (ANC) ≥ 1.0 x 109/L, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100 x 109/L.
12. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
13. Ejection fraction ≥ 50%, as measured by echocardiogram or multigated acquisition (MUGA) scan at Screening.
14. For women of childbearing potential (WCBP): negative serum beta human chorionic gonadotropin (betahCG) pregnancy test within 1 week before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months for women > 55 years of age).
15. Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study treatment, including 30 days after the last dose of SRF231. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception. Azoospermic males and WCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However female patients must still undergo pregnancy testing as described in this section.
16. Ability to adhere to the study visit schedule and all protocol requirements.
17. Signed and dated institutional review board (IRB)/independent ethics committee (IEC)-approved informed consent form before any screening procedures are performed.

Exclusion Criteria:

1. Previously received an anti-CD47 antibody or SIRPalpha targeted therapy.
2. High-grade lymphomas (eg, Burkitt's, lymphoblastic), plasma cell leukemia.
3. History of any condition known to be associated with reduced red blood cell (RBC) lifespan (eg, thalassemia trait, glucose-6-phosphate dehydrogenase deficiency).
4. History of ≥ Grade 4 allergic or anaphylactic reaction to any monoclonal antibody therapy, murine protein, or any excipient in the study drugs.
5. Major surgery within 4 weeks prior to Screening.
6. Symptomatic or untreated brain metastases (including leptomeningeal metastases).
7. Primary central nervous system malignancy.
8. Part A only: Prior RBC or platelet transfusion < 4 weeks prior to starting SRF231.
9. Prior autologous stem cell transplant ≤ 3 months prior to starting SRF231.
10. Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus.
11. Ongoing treatment with chronic immunosuppressants (eg, cyclosporine) or systemic steroids at doses used as anticancer therapy (ie, > 20 mg/day prednisone or equivalent) Note: topical, intranasal, or inhaled corticosteroids and physiologic replacement for patients with adrenal insufficiency are allowed.
12. Ongoing uncontrolled systemic bacterial, fungal, or viral infections at Screening Note: oral antibiotics for a controlled infection are permitted. Patients on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met.
13. Administration of a live vaccine within 6 weeks of first dose of study drug.
14. Prior allogeneic hematopoietic cell transplant within 6 months or with clinical Graft-Versus-Host Disease.
15. Previous chimeric antigen receptor (CAR)-T/T-cell receptor (TCR) cellular therapy with detectable circulating CAR-T/TCR cells.
16. History of autoimmune hemolytic anemia, autoimmune thrombocytopenia, atypical hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura.
17. Baseline QT interval corrected with Fridericia's method (QTcF) > 480 ms. Note: criterion does not apply to patients with a right or left bundle branch block.
18. Female patients who are pregnant or breastfeeding.
19. Concurrent active malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix.
20. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening.
21. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
[Part A] Dose-limiting toxicity (DLT) | Through 24 months with 21 day drug treatment cycles
  The number of patients in Part A who experienced a DLT during Cycle 1 or completed at least 75% of the prescribed Cycle 1 SRF231 dose will be used to assess tolerability and determine the appropriate dose for Part B.
[Part A] Non-tolerated Dose (NTD) | Through 24 months with 21 day drug treatment cycles
  For Part A, the NTD is the dose level at which 2 or more patients experience a DLT in the first cycle of treatment.
[Part A] Maximum tolerated Dose (MTD) | Through 24 months with 21 day drug treatment cycles
  For Part A, the MTD is defined as the dose level immediately below the non-tolerated dose (NTD). A total of 6 patients must be treated at a dose level for it to be considered the MTD.
[Parts A and B] Safety Analysis: summarizing adverse events (AEs) and will be based on treatment-emergent AEs (TEAEs) | Through 24 months with 21 day drug treatment cycles
  Safety and tolerability of SRF231 monotherapy will be assessed by summarizing adverse events (AEs) and will be based on treatment-emergent AEs (TEAEs). A TEAE is an AE that emerges or worsens in the period from the first dose of study treatment to 30 days after the last dose of study drug assessed by per CTCAE version 4.03 or higher.

SECONDARY OUTCOMES:
[Parts A and B] Maximum serum concentration (Cmax) of SRF231 | Up to 24 months
  Cmax in serum for all patients who receive at least one dose of SRF231 and had at least one measurable concentration based on the actual sample collection times determined using standard noncompartmental methods.
[Parts A and B] Time to maximum serum concentration (tmax) of SRF231 | Up to 24 months
  Tmax in serum for all patients who receive at least one dose of SRF231 and had at least one measurable concentration based on the actual sample collection times determined using standard noncompartmental methods.
[Parts A and B] Area under the serum concentration-time curve from time zero to the last quantifiable time point (AUC 0-last) of SRF231 | Up to 24 months
  AUC 0-last for all patients who receive at least one dose of SRF231 and had at least one measurable concentration based on the actual sample collection times determined using standard noncompartmental methods
[Parts A and B] Area under the serum concentration-time curve from time zero extrapolated to infinity (AUC 0-INF) of SRF231 | Up to 24 months
  AUC 0-INF for all patients who receive at least one dose of SRF231 and had at least one measurable concentration based on the actual sample collection times determined using standard noncompartmental methods.
[Parts A and B] Terminal elimination half-life (t1/2) of SRF231 | Up to 24 months
  T1/2 for all patients who receive at least one dose of SRF231 and had at least one measurable concentration based on the actual sample collection times determined using standard noncompartmental methods.
[Parts A and B] Pharmacodynamics of SRF231 via receptor occupancy | Up to 24 months
  Blood samples will be collected from all patients at multiple time points for analysis of CD47 receptor occupancy by SRF231. PD analyses will be descriptive and summary tabulations may be produced.
[Parts A and B] Anti-Drug Antibodies (ADAs). Time Frame: Up to 24 months | Up to 24 months
  Determine the incidence of ADAs in all patients who receive at least one dose of SRF231 and had at least one measurable sample.
[Part B] Overall Response Rate (ORR) including the best response of complete response (CR) or partial response (PR) | Up to 24 months
  ORR will be estimated by the percentage of patients achieving a best overall response of CR or PR using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, International Working Group Lugano Criteria (IWG Lugano) or other tumor-appropriate response criteria.
[Part B] Duration of Response (DOR) including time from the first documented to response to documented disease progression | Up to 24 months
  DoR defined as the time from first documented response to documented disease progression using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, International Working Group Lugano Criteria (IWG Lugano) or other tumor-appropriate response criteria will be summarized.
[Part B] Disease Control Rate (DCR) as the percentage of patients with CR, PR, or stable disease (SD) | Up to 24 months
  DCR defined as the percentage of patients with CR, PR or SD determined using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, International Working Group Lugano Criteria (IWG Lugano) or other tumor-appropriate response criteria will be summarized.
[Part B] Progression Free Survival as the time from first treatment to death or documented disease progression | Up to 24 months
  PFS defined as the time from the first treatment on study to death or documented disease progression using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, International Working Group Lugano Criteria (IWG Lugano) or other tumor-appropriate response criteria will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Study Chair — Surface Oncology
Locations (3):
- United States (2):
  - Research Site 002, New York, New York
  - Research Site 001, San Antonio, Texas
- Research Site 101, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No